CLINICAL TRIAL: NCT06544889
Title: A Single Center, Open-Label, Non-Randomized, Safety in Use Clinical Study to Assess The Topical Tolerability, Comedogenic and Acnegenic Potential, and Efficacy in Inflammatory and Non-Inflammatory Acne Vulgaris of a Sunscreen in Adult Subjects With Oily and Combination, Acne-Prone Skin
Brief Title: A Study to Assess the Safety and Efficacy of a Sunscreen on Acne-Prone Skin With Inflammatory and Non-Inflammatory Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JNTL Consumer Health (Brasil) LTDA (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS2024SK100019
Record Dates: First submitted 2024-08-05; First posted 2024-08-09 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sunscreen (Experimental): Eligible study participants will visit the Site for an initial evaluation of skin condition and receive the Sunscreen to be used at home. Next, participants will use the Sunscreen in normal conditions at home for 28 +/- 2 days, returning to the Site after 7 days of product use, then make the last study visit to complete the final analysis.
  Interventions: Other: Sunscreen SPF 70

INTERVENTIONS:
Other: Sunscreen SPF 70 — Participants will topically apply sunscreen SPF 70

SUMMARY:
The purpose of this trial is to evaluate 1) To assess the dermatological tolerability and the absence of acnegenic and comedogenic potential of 1 facial sunscreen, after 28 ± 2 days of use under normal conditions by adult subjects with acne prone skin, 2) To assess the clinical efficacy of the topical product in inflammatory and non-inflammatory acne vulgaris, and in the reduction of post-inflammatory erythema (PIE) and post-inflammatory hyperpigmentation (PIH) spots, under normal conditions of use; 3) Facial image capture with the VISIA-CR® Analysis System (Canfield Scientific, Inc.) equipment, to analyze acne marks and record before and after; 4)Assessment of perception by the study subject through Self-Perceived Effectiveness questionnaires and satisfaction surveys (emotional testimony).

ELIGIBILITY:
Inclusion Criteria:

* Men and/or Women;
* 18 to 55 years old;
* Subjects vaccinated against COVID-19;
* Subjects of all ethnicities according to IBGE criteria - IBGE-The Brazilian Institute of Geography and Statistics;
* Phototypes I to IV according to the Fitzpatrick classification;
* Oily or combination skin with a tendency to acne - confirmed by a dermatologist;
* Healthy skin in the test area (except for comedones and occasional inflammatory lesions - papules and pustules);
* Generally, in good health based on medical history reported by the subject;
* Subjects with mild elementary acne lesions (Grade 2 on the IGA scale), including non-inflammatory and/or inflammatory lesions (papules/pustules only, no nodular lesions) - proven by a dermatologist;
* Subjects presenting the following criteria on the face, confirmed by Expert Grader:

  1. At least 1 PIE
  2. At least PIH
* For male subjects: who agree to shave 24 hours before Visits 1, 2, and 3;
* Subjects able to read, write, speak, and understand Portuguese;
* Subjects who signed the terms ICD - Informed Consent Document and ICID - Informed Consent Image Disclosure;
* Intends to complete the study and is willing and able to follow all study instructions and attend the Site on the day(s) and at the time(s) set for the evaluations;

Exclusion Criteria:

* Has known allergies or adverse reactions to common topical skin care products including sunscreens; medications, or other products that the investigator deems relevant;
* Presents a skin condition that may confound the study results (specifically psoriasis, eczema, atopic dermatitis, cutaneous xerosis, erythema, or active skin cancer);
* Has self-reported Type 1 or Type 2 diabetes or is taking insulin or another anti-diabetic medication;
* Is taking a medication that would mask an Adverse Event (AE) or confound the study results, including:

  * Immunosuppressive or steroidal drugs within 2 months before Visit 1*
  * Non-steroidal anti-inflammatory drugs within 5 days before Visit 1* (For Oxaprozin and Piroxicam consider 2 weeks before visit 1).
  * Antihistamines within 2 weeks before Visit 1* *If an individual is taking one of these medication types, the individual is not considered eligible at screening. However, if a subject begins using one of these medications during the study, the Study Physician should be consulted to consider the impact of the specific medication on subject safety and/or the study results.
* Is currently using or has used any facial products containing acne active ingredients (e.g. benzoyl peroxide, salicylic acid, etc.) within the past 2 weeks or longer, if in the opinion of the Study Physician this could interfere with study results;
* Aesthetic or dermatologic treatment, invasive or non-invasive, in the test areas within 2 weeks prior to the start of the study and during the study;
* Subjects who reported being pregnant, or planning to become pregnant during the study;
* Using any medication to treat diseases of the face or eyes;
* Use of any other products capable of interfering with the study evaluations, at the discretion of the dermatologist;
* Subjects who have hormonal dysfunction that may influence the study results, at the discretion of the attending physician (for example, subjects with a history of irregular menstruation, polycystic ovary syndrome, users of anabolic steroids, and/or medication for hormone treatment, etc);
* Moderate to severe acne skin, confirmed by a dermatologist;
* Has a history of or a concurrent health condition/situation that may put the individual at significant risk, confound the study results, or interfere significantly with the individual's participation in the study;
* Has washed their face less than 2 hours before the study assessments;
* Excessive hair in the assessment area that could interfere with visual measurements. In the case of men, even in the presence of excessive hair in the beard area, they will be instructed to shave 24 hours before the visit;
* Simultaneously taking part in another study;
* Being an employee/contractor or close relative of the PI, Study Site, or Sponsor.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 28 days
  Number of participants with adverse events will be reported. An adverse event is any untoward medical occurrence in a clinical study participant temporally associated with the clinical investigation, whether or not the event has a causal relationship to the participants' participation in the trial. It is therefore any unfavorable and unintended sign (including an abnormal finding), symptom, or disease that occurs during the trial. This can include any occurrence that is new in onset, an aggravation of severity/frequency of a baseline condition, or abnormal results of diagnostic procedures, including laboratory test abnormalities.
Topical tolerability as assessed by the dermatologist | Baseline, Day 7 and Day 28 +/- 2 days
  Topical tolerability will be assessed using skin reaction intensity evaluation scale. Skin Reaction Intensity Evaluation Scale is a composite evaluation of any irritation/reaction subscoring for erythema, peeling, vesiculation, and edema. The scale ranges from 0=absent to 4=intense.
Number of Participants with Improvement from Baseline in Acne and Comedones | Baseline, Day 7 and Day 28 +/- 2 days
  The comedogenic and acnegenic potential will be evaluated by comparing the final acne lesion counts (D28) with the baseline acne lesion counts. The lesions will be classified as closed comedones (whiteheads), open comedones (blackheads), pustules (pustules) and papules (papules). The lesions will be counted in 05 areas of the face: 02 in the frontal region, 02 in the malar region and chin, papules and pustules will be counted on the entire face (except the nose).
Change from Baseline in Clinical Effectiveness Assessment on Post-Inflammatory Hyperpigmentation | Baseline, Day 7 and Day 28 +/- 2 days
  Change from Baseline in Clinical Effectiveness Assessment on Post-Inflammatory Hyperpigmentation (PIH) will be reported. A 10-point ordinal scale (0 to 9) will be used. Therefore, as it is an ordinal scale, the intermediate points do not have an established definition. For PIH, the evaluated area will be the Global Face and the scale to be used is defined from 0 = None, uniform skin color with no observable hyperpigmentation to 9 = Severe/highly visible, deep color difference.
Change from Baseline in Clinical Effectiveness Assessment on Post-Inflammatory Erythema | Baseline, Day 7 and Day 28 +/- 2 days
  Change from Baseline in Clinical Effectiveness Assessment on Post-Inflammatory Erythema (PIE) will be reported. A 10-point ordinal scale (0 to 9) will be used. Therefore, as it is an ordinal scale, the intermediate points do not have an established definition. For PIE, the evaluated area will be the Global Face and the scale to be used is defined from 0 = None, skin color without observable erythema to 9 = Severe/Highly visible, color difference between skin and spot intense.
Number of Participants with Improvement From Baseline in Acne Mark Attributes Assessed Using the Visia-CR Facial Imaging Booth | Baseline, Day 7 and Day 28 +/- 2 days
  Facial images will be captured using the Visia CR Facial Imaging Booth. Three Three images per participant will be captured: right lateral, left lateral and frontal using using the Cross Polarized, Standard 2 and RBX (Red) filters. The captured images will be further analyzed using specific image analysis software to evaluate the reduction in acne, improvement in PIE and PIH, reduction in acne marks.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 7 | Day 7
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 7 will be reported. Participants will answer 11 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.
Participant's Self-perceived Questionnaire to Assess the Clinical Effectiveness of the Sunscreen on Day 28 | Day 28 +/- 2 days
  Participant's self-perceived questionnaire to assess the clinical effectiveness of the sunscreen on Day 28 will be reported. Participants will answer 11 questions and rate as: totally disagree, disagree, neither agree nor disagree, agree and totally agree.
Testimonial Regarding the Experience with Sunscreen | End of the study (Day 28 +/- 2 days)
  A testimonial regarding the experience with sunscreen will be provided by the participants through an open question at the end of the study. The purpose is to know their opinion and experience using this product during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielli Brianezi, PhD, Principal Investigator — Johnson & Johnson Consumer Inc. (J&JCI)
Locations (1):
- Allergisa Pesquisa Dermato-Cosmética Ltda, Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No